CLINICAL TRIAL: NCT02485028
Title: An Open Label, Randomized, Single-dose Crossover Study to Evaluate the Pharmacokinetic Interaction of Dapoxetine 30mg and Mirodenafil 50mg in Healthy Male Volunteers
Brief Title: Pharmacokinetic Interaction Study of Dapoxetine 30mg and Mirodenafil 50mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SID123_DDI_I_2013; 12542 (Other: South Korea: Ministry of Food and Drug Safety)
Record Dates: First submitted 2015-06-10; First posted 2015-06-30 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Drug Interaction Potentiation
Keywords: Dapoxetine; Mirodenafil; DDI study
MeSH Terms: interventions — dapoxetine; Tablets; mirodenafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- M→D→D+M (Experimental): Mirodenafil(M) in period 1, Dapoxetine(D) in period 2, Dapoxetine+Mirodenafil(D+M) in period 3
  Interventions: Drug: Dapoxetine 30mg tablet; Drug: Mirodenafil 50mg tablet
- M→D+M→D (Experimental): Mirodenafil(M) in period 1, Dapoxetine+Mirodenafil(D+M) in period 2, Dapoxetine(D) in period 3
  Interventions: Drug: Dapoxetine 30mg tablet; Drug: Mirodenafil 50mg tablet
- D→M→D+M (Experimental): Dapoxetine(D) in period 1, Mirodenafil(M) in period 2, Dapoxetine+Mirodenafil(D+M) in period 3
  Interventions: Drug: Dapoxetine 30mg tablet; Drug: Mirodenafil 50mg tablet
- D+M→M→D (Experimental): Dapoxetine+Mirodenafil(D+M) in period 1, Mirodenafil(M) in period 2, Dapoxetine(D) in period 3
  Interventions: Drug: Dapoxetine 30mg tablet; Drug: Mirodenafil 50mg tablet
- D+M→D→M (Experimental): Dapoxetine+Mirodenafil(D+M) in period 1, Dapoxetine(D) in period 2, Mirodenafil(M) in period 3
  Interventions: Drug: Dapoxetine 30mg tablet; Drug: Mirodenafil 50mg tablet
- D→D+M→M (Experimental): Dapoxetine(D) in period 1, Dapoxetine+Mirodenafil(D+M) in period 2, Mirodenafil(M) in period 3
  Interventions: Drug: Dapoxetine 30mg tablet; Drug: Mirodenafil 50mg tablet

INTERVENTIONS:
Drug: Dapoxetine 30mg tablet
Drug: Mirodenafil 50mg tablet

SUMMARY:
Healthy male volunteers were administered alone and in combination with dapoxetine 30mg mirodenafil 50mg for three times, respectively and the pharmacokinetic interaction was compared between the two drugs.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male adults aged between 19 and 55
* Body mass index (BMI) in the range of 19 to 27 kg/m2
* Understand the requirements of the study and voluntarily consent to participate in the study
* Available for the entire study period

Exclusion Criteria:

* Subject has a history such as liver diseases, kidneys, digestive system, respiratory system, endocrine system, nervous psychiatric, blood, cancer, cardiovascular diseases
* Subject with clinically significant vital signs (sitting position blood pressure) (90 mmHg > systolic blood pressure ≥ 140 mmHg, 60 mmHg > diastolic blood pressure ≥ 90 mmHg)
* History of drug abuse
* History of caffeine, alcohol, smoking abuse

  * caffeine(coffee,tea,coke)> 4cups/day
  * smoking > 10 cigarettes/day
  * alcohol > 140g/week
* Consumption of any grapefruit or grapefruit-containing juices over 1 cup a day
* Previously donate whole blood within 60 days or component blood within 30 days
* Subject has taken drugs which affects the ADME of investigational products
* Subject with known for hypersensitivity reactions to mirodenafil/ dapoxetine or other drugs
* Inadequate laboratory test result:

  * AST(SGOT) or ALT(SGPT) or total bilirubin > 1.5 x upper limit of normal range
  * eGFR < lower limit of normal range
* Subject considered as unsuitable based on medical judgement by investigators

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Cmax | predose, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours post-dose
  Cmax of dapoxetine and mirodenafil
Area Under Curve (AUC) | predose, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours post-dose
  AUC of dapoxetine and mirodenafil

SECONDARY OUTCOMES:
Tmax | predose, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours post-dose
t1/2 | predose, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours post-dose
CL/F | predose, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours post-dose
Vd/F | predose, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours post-dose
Number of Participants with Adverse Events | During 22 days from first administration of period 1
  Incidence rate of Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Wook Ko, MD, PhD, Principal Investigator — Samsung Medical Center